CLINICAL TRIAL: NCT06612138
Title: Pilates, Yoga and Tai Chi Exercises' Effect on Balance and Gait in Patients With Multiple Sclerosis
Acronym: MS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, principal investigator: alshaymaa shaaban abd el azeim, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005332
Record Dates: First submitted 2024-09-21; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Multiple Sclerosis
Keywords: pilates; yoga; tai chi; multiple scelerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: pilates, yoga, tai chi and traditional therapy
Who Masked: Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pilates exercises (Experimental): the patients will receive pilates exercise twice a week for six weeks plus traditional
  Interventions: Other: pilates exercises; Other: tradional physical therapy
- yoga exercise (Experimental): the patients will receive yoga exercise twice a week for six weeks plus traditional
  Interventions: Other: yoga exercises; Other: tradional physical therapy
- tai chi exercises (Experimental): the patients will receive tai chi exercise twice a week for six weeks plus traditional
  Interventions: Other: tai chi exercises; Other: tradional physical therapy
- traditional physical therapy (Active Comparator): the patients will receive tradional physical therapy twice a week for six weeks
  Interventions: Other: tradional physical therapy

INTERVENTIONS:
Other: pilates exercises — the patients will receive pilates exercises in the form of breathing exercises, chest lift, bridging, mermaid, swan, quadruped exercises
  Arms: Pilates exercises
Other: yoga exercises — the patients will receive yoga in the form of Bhastrikā: rapid and powerful inhalations and exhalations by means of the force of the diaphragm, letting the air sound when exhaling, Nāḏī Śoḏhana: from Sanskrit, "nadi" means 'to channel' and "shodhana" means 'purify, cleanse', o Hand position "Mrigi mudra": It consists of flexing the index and ring fingers of the hand, o Breathing: Gently close the right nostril with the thumb, inhale fingers and exhale slowly through the right. Keeping your right nostril open, inhale, close it, and slowly open and exhale through the left. This is a cycle. Repeat 3-5 times and then release the hand mudra and return to normal breathing.
  Arms: yoga exercise
Other: tai chi exercises — the patients will receive tai chi in the form of Commencing form, Repulse Monkey,Grasp Peacock's Tail,Move Hands like Moving Clouds (left side only), Fair Lady Works at Shuttles, Golden Cock Stands on One Leg (left and right),Brush Knees and Twist Steps, Closing form.
  Arms: tai chi exercises
Other: tradional physical therapy — Patients will receive traditional physiotherapy breathing, massage and relaxation exercises

SUMMARY:
this study will be conducted to compare between the effect of Pilates, Yoga and Tai Chi on balance, gait ability, functional mobility and fatigue in patients with multiple sclerosis

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic immune-mediated disease involving inflammation, plaques, and demyelination in the central nervous system . MS typically affects people in early adulthood in the 20-40 year range and is two to three times more common in women than men. Exercise therapy is one of the greatest and most well-researched rehabilitation strategies for multiple sclerosis patients. Exercise therapy includes a variety of exercise methods, including resistance training and endurance training, all of which are suitable for multiple sclerosis patients to use. Exercise can alter a wide range of functional and health-related factors as well as the diversity of symptoms displayed by multiple sclerosis patients.Pilates is a method of physical exercise that focuses on core stability, strength, flexibility, posture, muscle control, breathing, and mind-body connection.Yoga therapy is the process of empowering individuals to progress toward improved health and well-being through the application of the philosophy and practice of Yoga. Practicing yoga can provide the tools to help patients with multiple sclerosis cope with the disease and manage everyday tasks in a more beneficial way .Tai Chi is a martial art of Chinese origin that is based on the development of inner energy by practicing predetermined movements softly. It is an intense and complete practice, beneficial at any age. Tai Chi thus falls within a long tradition in Chinese therapies and exercises to improve the individuals' quality of life. 100 patients with multiple sclerosis will be allocated randomly to four groups; group1 will receive pilates plus traditional therapy, group 2 will receive yoga plus traditional therapy, group 3 will receive tai chi plus traditional therapy and group 4 will receive traditional therapy only.

ELIGIBILITY:
Inclusion Criteria:

* A score of 3.5 or less on the Expanded Disability Status Scale (EDSS) because individuals with an EDSS score greater than 3.5 need more assistance, being less independent (Zorina et al.,2020).
* All patients are taking their conventional medical treatment of relapsing-remitting stage
* Age over than 18 years
* All definite multiple sclerosis patients diagnosed as MS according to revised McDonald criteria 2017 .
* Both males and females will be included
* All Patients will be referred from neurologist.

Exclusion Criteria:

Patients will be excluded if their diagnosis is not clearly established, if they suffer from an acute relapse or severe cognitive deficits, or have signs of any psychiatric disease -Brain surgery/trauma/history of brain disease (stroke), other independent neurological history

* Another exclusion criterion is the history of cardiac, pulmonary, orthopedic,or other medical conditions diagnosed before participation
* Rheumatic diseases and other acute or chronic inflammations
* Vascular disease, spinal cord compression, vitamin B 12 deficiency
* Other conditions that affect the smooth progress of the inspection: such as hearing impairment, comprehension impairment, poor compliance
* Alcoholism or drug dependence (addiction)
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
balance | up to six weeks
  The Berg Balance Scale (BBS) was developed to measure balance. The BBS consists of 14 functional balance items.Each item is scored on a 5-point ordinal scale ranging from 0 to 4, with 0 indicating an inability to complete the task entirely and 4 indicating an ability to complete the task criterion.A score of 56 indicates functional balance; and scores below 45 indicate greater risk for falling.
gait assessment | up to six weeks
  12-Item Multiple Sclerosis Walking Scale is valid and reliable to assess gait ability in patients with multiple sclerosis. Patients are asked to answer 12 questions about limitations to their walking due to MS over the past 2 weeks, circling a number that best describes their degree of restriction (1, not at all; 2, a little; 3, moderately; 4, quite a bit; 5, extremely). Higher scores indicate the higher impact of the disease on walking. Finally, the score of walking ability falls into a 48-point range with minimum and maximum scores of 12 and 60.
exercise capacity | up to six weeks
  6 Minute Walk Test is valid and reliable for the evaluation of exercise capacity.The patient is instructed to 'walk at your comfortable pace' back and forth along a hallway for 6 minutes. The maximum distance walked is measured and recorded

SECONDARY OUTCOMES:
functional mobility | up to six weeks
  Timed up and go test (TUG) is valid and reliable for the evaluation of functional mobility in patients with multiple sclerosis.A score of ≥ 14 seconds has been shown to indicate high risk of fall, while score ≤10 seconds = normal, score ≤ 20 seconds = good mobility, can go out alone, mobile without gait aid, score ≤ 30 seconds = problems and cannot go outside alone and requires gait aid
fatigue | up to six weeks
  The Fatigue Severity Scale (FSS), originally developed by Krupp for use in patients with MS, has been used to measure fatigue. It consists of 9 items.patients score each item from 1 to 7, based on the extent, to which they agree or disagree with each statement (1 = strong disagreement, 7 = strong agreement). The FSS can be scored either by obtaining a total score, or by calculating a mean score across all 9 items, with higher scores indicating more severe fatigue
life disability | up to six weeks
  Multiple sclerosis quality of life questionnaire will be used to assess life disability. MSQoL-54 scale scores were created using the Likert method by averaging items within the scales and, then row scores were linearly transformed into 0-100 scales. Higher values indicate better quality of life.